CLINICAL TRIAL: NCT04639544
Title: Randomized, Triple-blind, Parallel-group Study to Evaluate the Effect of Consuming a Lactobacillus Strain on the Prevention of Recurrent Vaginal Candidiasis
Brief Title: Effect of a Lactobacillus Strain on the Prevention of Recurrent Vaginal Candidiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P049
Record Dates: First submitted 2020-10-16; First posted 2020-11-20 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Recurrent Vulvovaginal Candidiasis
Keywords: Recurrent Vulvovaginal Candidiasis; Prevention; Probiotics
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Volunteers will take 1 capsule per day with maltodextrin for 6 months
  Interventions: Dietary Supplement: Placebo
- Probiotic group (Experimental): Volunteers will take 1 capsule per day with the Lactobacillus strain for 6 months
  Interventions: Dietary Supplement: Lactobacillus strain

INTERVENTIONS:
Dietary Supplement: Placebo — Each participant will consume 1 capsule per day in one of the main meals without any restriction in the diet or in their life habits
  Arms: Control group
Dietary Supplement: Lactobacillus strain — Each participant will consume 1 capsule per day in one of the main meals without any restriction in the diet or in their life habits
  Arms: Probiotic group

SUMMARY:
The objective of this study is to evaluate the efficacy of the consumption of the one probiotic strain in the prevention of new vaginal candidiasis events in women with recurrent vaginal candidiasis. This is a preliminary study whose purpose is to know if this probiotic is effective in reducing the number of candidiasis events and / or increasing the time between possible relapses in women diagnosed with RVVC.

DETAILED DESCRIPTION:
Previous studies have demonstrated the effectiveness of certain probiotic strains in the treatment of vaginal candidiasis, alone or as an adjunct to antifungal treatments, as well as the effectiveness of a Lactobacillus strain as maintenance treatment after antifungal treatment to reduce the recurrence rate of candidiasis However, to date, no studies have evaluated the oral efficacy of a probiotic strain of Lactobacillus originally isolated from breast milk in the prevention of new vaginal yeast events in women with recurrent vaginal yeast infections.

The objective of this study is to evaluate the efficacy of the consumption of the one probiotic strain in the prevention of new vaginal candidiasis events in women with recurrent vaginal candidiasis. This is a preliminary study whose purpose is to know if this probiotic is effective in reducing the number of candidiasis events and / or increasing the time between possible relapses in women diagnosed with RVVC.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women from 18 to 49 years old.
2. Having suffered at least four outbreaks of vaginal yeast infection in the last year.
3. Signed Informed Consent Form.
4. Agree to provide the scheduled samples.
5. Agree to perform gynecological examinations
6. Agree to report candidiasis events that occur during the study.
7. Ability to complete surveys.

Exclusion Criteria:

1. Being currently consuming or having consumed a probiotic in the two weeks prior to the study.
2. Being under antibiotic treatment at the time of beginning the study.
3. Being under pharmacological treatment for the treatment of candidiasis.
4. Have an allergy to an antibiotic

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of candidiasis events | 6 months
  Total candidiasis events during intervention
Time between episodes | 6 months
  Days from baseline until candidiasis events

SECONDARY OUTCOMES:
Determination of Candida in vaginal exudate by culture analysis | 6 months
  Analysis of the presence of Candida in vaginal exudate
Microbiota of vaginal exudate | 6 months
  Load of Candida, Lactobacillus, Gardnerella, Prevotella, Streptococcus and Bacteroides species in vaginal exudate samples
Gynecological examination | 6 months
  The gynecologist will perform a gynecological examination to check:Presence of erythema of the vulva, erythema of the vaginal mucosa, lumpy, whitish-coloured vulvar oedema and excoriation of the vulva
pH of vaginal discharge | 6 months
  Measurement of the pH of vaginal discharge
Test of related clinical symptoms | 6 months
  The volunteers will complete a test about presence of vaginal itching, vaginal burning, whitish vaginal discharge, dysuria and dyspareunia.
Intensity of the related clinical symptoms | 6 months
  Intensity (mild, moderate, intense) of the related clinical symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jose Maldonado Lobón, PhD, Principal Investigator — Biosearch S.A.
Locations (1):
- Hospital Universitario Infanta Elena, Valdemoro, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No